CLINICAL TRIAL: NCT04737915
Title: Comparing the Efficacy of a Single-Session Virtual Reality Treatment for Fear of Heights to In Vivo Exposure and No Treatment
Brief Title: Virtual Reality Exposure Versus In Vivo Exposure for Fear of Heights
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Notre Dame (Other)
Responsible Party: Principal Investigator, Jennifer Hames, Assistant Clinical Professor & Clinic Director, University of Notre Dame
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Interventional
Record Dates: First submitted 2021-01-28; First posted 2021-02-04 (Actual); Last update posted 2021-02-08 (Actual); Status verified 2021-02

CONDITIONS: Fear of Heights; Acrophobia; Specific Phobia; Anxiety Disorder
MeSH Terms: conditions — Acrophobia; Phobia, Specific; Anxiety Disorders | interventions — Implosive Therapy; Virtual Reality Exposure Therapy

STUDY DESIGN:
Intervention Model Description: Eligible participants were randomly assigned to one of three conditions: a) single session virtual reality exposure; b) single session in vivo exposure; c) waitlist control
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Virtual Reality Exposure (Experimental): Participants completed a single session of exposure administered via a virtual reality headset. The exposure exercise involved looking over virtual railings into an atrium at various floor levels (the virtual environment was designed to look like the atrium in the in vivo exposure condition). Exposure was conducted in six 6-minute trials for a total of 36 minutes of exposure.
  Interventions: Behavioral: Exposure Therapy (Virtual Reality)
- In Vivo Exposure (Experimental): Participants completed a single session of exposure administered in vivo. The exposure exercise involved looking over actual railings into an atrium at various floor levels. Exposure was conducted in six 6-minute trials for a total of 36 minutes of exposure.
  Interventions: Behavioral: Exposure Therapy (In Vivo)
- Waitlist Control (No Intervention): Participants watched a neutral video during the time participants in other conditions were completing the exposure exercise. Participants received no exposure-based intervention.

INTERVENTIONS:
Behavioral: Exposure Therapy (In Vivo) — Participant completes a single session of exposure therapy for fear of heights by looking over railings into an atrium at various floor levels in a virtual environment.
  Arms: In Vivo Exposure
Behavioral: Exposure Therapy (Virtual Reality) — Participant completes a single session of exposure therapy for fear of heights by looking over railings into an atrium at various floor levels in a real environment.
  Arms: Virtual Reality Exposure

SUMMARY:
This study randomly assigned 114 participants with significant fear of heights to one of three conditions: a) a single session of virtual reality exposure; b) a single session of in vivo exposure; or c) a control condition. The aim of this study was to compare the efficacy of virtual reality exposure to the efficacy of in vivo exposure or no exposure for participants with significant fear of heights.

ELIGIBILITY:
Inclusion Criteria:

* Score >= 45 on the Acrophobia Questionnaire (AQ)

Exclusion Criteria:

* Already receiving therapy specifically for fear of heights.
* Has any contraindications to using a virtual reality headset.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2018-06-11 (Actual); Primary Completion 2019-03-06 (Actual); Study Completion 2019-03-06 (Actual)

PRIMARY OUTCOMES:
Acrophobia Questionnaire (AQ) | Immediately Post-Treatment (Controlling for Baseline Scores)
  Participants completed the anxiety subscale of the AQ, a 20-item questionnaire that assesses self-reported anxiety related to acrophobia. Scores for the subscale are summed, and totals range from 0 to 120, with higher scores indicating greater anxiety.
Behavioral Approach Task (BAT) | Immediately Post-Treatment (Controlling for Baseline Scores)
  Participants walked up a staircase until they reach the highest level they can complete, while stopping to look over the ledge toward the floor at each landing. During each BAT, fear response was assessed behaviorally (highest step reached) and subjectively (self reported levels of fear).
Heights Interpretation Questionnaire (HIQ) | Immediately Post-Treatment (Controlling for Baseline Scores)
  Participants completed the HIQ, a 16-item questionnaire that assesses self-reported interpretations of an imagined experience of heights. Items are summed scored, and totals ranged from 16 to 80, with higher scores indicating greater height fear-relevant interpretation bias.
Acrophobia Questionnaire (AQ) | 1-Week Post-Treatment (Controlling for Immediate Post-Treatment Scores)
  Participants completed the anxiety subscale of the AQ, a 20-item questionnaire that assesses self-reported anxiety related to acrophobia. Scores for the subscale are summed, and totals range from 0 to 120, with higher scores indicating greater anxiety.
Behavioral Approach Task (BAT) | 1-Week Post-Treatment (Controlling for Immediate Post-Treatment Scores)
  Participants walked up a staircase until they reach the highest level they can complete, while stopping to look over the ledge toward the floor at each landing. During each BAT, fear response was assessed behaviorally (highest step reached) and subjectively (self reported levels of fear).
Heights Interpretation Questionnaire (HIQ) | 1-Week Post-Treatment (Controlling for Immediate Post-Treatment Scores)
  Participants completed the HIQ, a 16-item questionnaire that assesses self-reported interpretations of an imagined experience of heights. Items are summed scored, and totals ranged from 16 to 80, with higher scores indicating greater height fear-relevant interpretation bias.

OTHER OUTCOMES:
Anxiety Sensitivity Index (ASI) | Baseline, Immediately Post-Treatment; 1 Week Post-Treatment
  The ASI is a 16 item measure assessing participants' fear of and sensitivity to physiological symptoms of anxiety. Scores range from 0-64, with higher scores indicating higher levels of anxiety sensitivity.
Affective Control Scale (ACS) - Anxiety Subscale | Baseline, Immediately Post-Treatment; 1 Week Post-Treatment
  The 13-item anxiety subscale of the ACS measures participants' fear tolerance. Scores range from 13-91, with higher scores indicating lower levels of anxiety fear tolerance.
High Place Phenomenon Index (HPPI) | Baseline, Immediately Post-Treatment; 1 Week Post-Treatment
  The HPPI is a 3-item measure that assesses participants' self-reported experience of the high place phenomenon. Scores range from 3-21, with higher scores indicating more frequent experience of the high place phenomenon.
Patient Health Questionnaire (PHQ) - 8 item version | Baseline, Immediately Post-Treatment; 1 Week Post-Treatment
  The PHQ is traditionally a 9 item measure, but this study used an 8 item version that did not include item 9 (assessing suicidality). Scores on this version range from 0 to 24, with higher scores indicating higher levels of depressive symptoms.
DSM-5 (Diagnostic and Statistical Manual of Mental Disorders - 5) Severity Measure for Specific Phobia (Adapted for Acrophobia) | Baseline, Immediately Post-Treatment; 1 Week Post-Treatment
  Participants completed the DSM-5 Severity Measure, a 10-item questionnaire that assesses the severity of DSM-5 symptoms of specific phobias. Total scores range from 0 to 40, with higher scores indicating higher levels of specific phobia symptomology.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer L Hames, Ph.D., Principal Investigator — University of Notre Dame
Locations (1):
- University of Notre Dame, Notre Dame, Indiana, United States

IPD SHARING:
Plan to Share IPD: No
Study protocols and de-identified data will be shared at the request of other researchers.